CLINICAL TRIAL: NCT00692718
Title: N-3 Fatty Acids for the Prevention of Atrial Fibrillation in Patients With Acute Heart Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Osaka General Medical Center (Other)
Responsible Party: Masaharu Masuda, Osaka Geneeal Medical Cener
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OFAHeft
Record Dates: First submitted 2008-05-29; First posted 2008-06-06 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Acute Heart Failure; Acute Myocardial Infarction
MeSH Terms: interventions — eicosapentaenoic acid ethyl ester; Eicosapentaenoic Acid

INTERVENTIONS:
Drug: Epadel, Eicosapentaenoic acid — Epadel 900mg, 2 times a day, during hospitalization

SUMMARY:
Our study is to investigate the effect of N-3 Fatty Acids for the prevention of atrial fibrillation in patients with acute heart failure or acute myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

* sinus rhythm patients with acute heart failure or acute myocardial infarction

Exclusion Criteria:

* pregnancy,allergy to epadel

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
detection of atrial fibrillation on ECG monitoring | anytime during hospitalization